CLINICAL TRIAL: NCT03402451
Title: Korean Stroke Cohort for Functioning and Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2012-06-016-001
Record Dates: First submitted 2018-01-01; First posted 2018-01-18 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Stroke; Disability; Function; Rehabilitation; Burden
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Korean Stroke Cohort for functioning and rehabilitation (KOSCO) is a large, multi-centre prospective cohort study for all acute first-ever stroke patients admitted to participating hospitals in nine distinct areas of Korea. This study is designed as a 10-year, longitudinal follow-up investigating the residual disabilities, activity limitations, and quality of life issues arising in patients suffering from first-ever stroke. The main objectives of this study are to identify the factors that influence residual disability and long-term quality of life. The secondary objectives of this study are to determine the risk of mortality and recurrent vascular events in patients with acute first-ever stroke. Investigators will investigate longitudinal health behaviors and patterns of healthcare utilization, including stroke rehabilitation care. Investigators will also investigate the long-term health status, mood, and quality of life in stroke patient caregivers. In addition, investigators will identify baseline and ongoing characteristics that are associated with secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. First-ever acute stroke (ischemic stroke or intracerebral hemorrhage) with corresponding lesion and/or evidence of acute arterial occlusion on CT (A)- or MRI/A-scan.
2. Age ≥ 19 years at onset of stroke.
3. Onset of symptoms within seven days prior to inclusion.

Exclusion Criteria:

1. Transient ischemic attack.
2. History of stroke.
3. Traumatic intracerebral hemorrhage.
4. Not Korean.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with an acute first-ever stroke, admitted to the representative hospitals in the nine distinct areas of Korea, will be asked to participate in the study. Participating study centres are Samsung Medical Center, Seoul; Severance Hospital, Seoul; Konkuk University Hospital, Seoul; Chungnam National University Hospital, Daejeon; Chonnam National University Hospital, Gwangu; Pusan National University Yangsan Hospital, Yangsan; Kyungpook National University Hospital, Deagu; Wonkwang University Hospital, Iksan; and Jeju National University Hospital, Jeju.
Sampling Method: Non-Probability Sample
Enrollment: 7858 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Korean modified Barthel Index | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for activities of daily living
Change in Euro Quality of Life-5 Dimensions | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for quality of life
Change in Functional Independence Measurement | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for activities of daily living
Change in Korean Mini-Mental State Examination | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for cognitive function
Change in Korean Version of Frenchay Aphasia Screening Test | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for language function
Change in modified Rankin Scale | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  Measurement for disability. Range of total score 0 to 6. 0 is no disability at all and 6 is death. Therefore, greater value means worse functional status
Change in American Speech-Language-Hearing Association National Outcome Measurement System Swallowing Scale | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  Measurement for swallowing function. Range of scale is 0 to 7, and greater value means better function. For example, 7 means no swallowing difficulty at all.
Change in Geriatric depression scale-short form | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for depression. The scale is 0 to 15. 0 is normal whereas 15 indicates severe depression.
Change in Fugl-Meyer Assessment | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for motor function
Change in Functional Ambulatory Category | 7 days, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months after stroke onset
  measurement for gait function

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang WH, Sohn MK, Lee J, Kim DY, Lee SG, Shin YI, Oh GJ, Lee YS, Joo MC, Han EY, Kim YH. Korean Stroke Cohort for functioning and rehabilitation (KOSCO): study rationale and protocol of a multi-centre prospective cohort study. BMC Neurol. 2015 Mar 25;15:42. doi: 10.1186/s12883-015-0293-5. PMID 25886039
- [Result] Chang WH, Sohn MK, Lee J, Kim DY, Lee SG, Shin YI, Oh GJ, Lee YS, Joo MC, Han EY, Kang C, Kim YH. Predictors of functional level and quality of life at 6 months after a first-ever stroke: the KOSCO study. J Neurol. 2016 Jun;263(6):1166-77. doi: 10.1007/s00415-016-8119-y. Epub 2016 Apr 25. PMID 27113602
- [Result] Yoon JA, Kim DY, Sohn MK, Lee J, Lee SG, Lee YS, Han EY, Joo MC, Oh GJ, Han J, Park M, Park KP, Noh KH, Chang WH, Shin YI, Kim YH. Factors associated with improvement or decline in cognitive function after an ischemic stroke in Korea: the Korean stroke cohort for functioning and rehabilitation (KOSCO) study. BMC Neurol. 2017 Jan 10;17(1):9. doi: 10.1186/s12883-016-0780-3. PMID 28073355
- [Result] Chang WH, Sohn MK, Lee J, Kim DY, Lee SG, Shin YI, Oh GJ, Lee YS, Joo MC, Han EY, Kim MS, Jang SY, Kim JH, Kim YH. Long-term functional outcomes of patients with very mild stroke: does a NIHSS score of 0 mean no disability? An interim analysis of the KOSCO study. Disabil Rehabil. 2017 May;39(9):904-910. doi: 10.3109/09638288.2016.1170214. Epub 2016 May 20. PMID 27206550
- [Result] Chang WH, Sohn MK, Lee J, Kim DY, Lee SG, Shin YI, Oh GJ, Lee YS, Joo MC, Han EY, Kim JH, Kim YH. Return to work after stroke: The KOSCO Study. J Rehabil Med. 2016 Mar;48(3):273-9. doi: 10.2340/16501977-2053. PMID 26843361
- [Result] Jang SY, Sohn MK, Lee J, Kim DY, Lee SG, Shin YI, Oh GJ, Lee YS, Joo MC, Han EY, Chang WH, Lee A, Kim JH, Kim YH. Chronic Kidney Disease and Functional Outcomes 6 Months after Ischemic Stroke: A Prospective Multicenter Study. Neuroepidemiology. 2016;46(1):24-30. doi: 10.1159/000441281. Epub 2015 Nov 26. PMID 26606379
- [Result] Yoon JA, Kim DY, Sohn MK, Lee J, Lee SG, Lee YS, Han EY, Joo MC, Oh GJ, Han J, Lee SW, Park M, Chang WH, Shin YI, Kim YH. Effect of stress hyperglycemia and intensive rehabilitation therapy in non-diabetic hemorrhagic stroke: Korean Stroke Cohort for Functioning and Rehabilitation. Eur J Neurol. 2016 Nov;23(11):1658-1665. doi: 10.1111/ene.13101. Epub 2016 Jul 22. PMID 27444813
- [Result] Jang SY, Shin YI, Kim DY, Sohn MK, Lee J, Lee SG, Oh GJ, Lee YS, Joo MC, Han EY, Chang WH, Kang C, Kim YH. Effect of obesity on functional outcomes at 6 months post-stroke among elderly Koreans: a prospective multicentre study. BMJ Open. 2015 Dec 18;5(12):e008712. doi: 10.1136/bmjopen-2015-008712. PMID 26685024
- [Derived] Shin M, Sohn MK, Lee J, Kim DY, Lee SG, Shin YI, Oh GJ, Lee YS, Joo MC, Han EY, Han J, Ahn J, Chang WH, Shin MA, Choi JY, Kang SH, Kim Y, Kim YH. Effect of Cognitive Reserve on Risk of Cognitive Impairment and Recovery After Stroke: The KOSCO Study. Stroke. 2020 Jan;51(1):99-107. doi: 10.1161/STROKEAHA.119.026829. Epub 2019 Dec 11. PMID 31822247
- [Derived] Han J, Lee HI, Shin YI, Son JH, Kim SY, Kim DY, Sohn MK, Lee J, Lee SG, Oh GJ, Lee YS, Joo MC, Han EY, Chang WH, Kim YH. Factors influencing return to work after stroke: the Korean Stroke Cohort for Functioning and Rehabilitation (KOSCO) Study. BMJ Open. 2019 Jul 11;9(7):e028673. doi: 10.1136/bmjopen-2018-028673. PMID 31300502